CLINICAL TRIAL: NCT04133701
Title: The Impact of Meal Timing on Neurovascular Control in Adults
Brief Title: Meal Timing and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-0417; A176000 (Other: UW Madison); EDUC/KINESIOLOGY/KINESIO (Other: UW Madison); Protocol Version 5/4/2021 (Other: UW Madison)
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Blood Pressure; Neurovascular Control
Keywords: Meal Timing; Blood Pressure; Time-Restricted Feeding; Sympathetic Nerve Activity
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: The interventional study model used will consist of a time-restricted feeding intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time-Restricted Feeding (Experimental): Control (Baseline): Blood pressure and neurovascular control will be measured.
  Post-Intervention: Blood pressure and neurovascular control will be measured.
  Interventions: Behavioral: Time-Restricted Feeding

INTERVENTIONS:
Behavioral: Time-Restricted Feeding — After baseline measurements have been completed, participants will enroll in a time-restricted feeding intervention. Participants will be asked to restrict the time in which they eat each day to 10 hours, fasting for the remaining 14 hours. Participants will also be asked to finish their last meal of the day at least 2 hours prior to bedtime.

SUMMARY:
Brain blood flow, blood pressure, and neurovascular control mechanisms will be measured in middle-aged adults before and after a brief intervention period. The intervention will consist of changing the time in which the participant consumes food each day.

DETAILED DESCRIPTION:
Healthy adults experience a 10-20% decrease in night-time blood pressure, compared with day-time blood pressure. However, 20-40% of middle-aged adults do not demonstrate a decrease in blood pressure. Abnormal blood pressure patterns are linked to sleep disturbances, hypertension, and associated with elevated cardiovascular risk and mortality. Additionally, abnormal diurnal blood pressure patterns are associated with impaired neurovascular control of the circulation, contributing to an increased risk of hypertension, stroke, and cardiovascular disease. Importantly, midlife is the critical period for implementing interventions to prevent or delay future cardiovascular disease. Recent data demonstrates that time-restricted feeding may normalize blood pressure patterns. The overall goal of this study is to determine if time-restricted feeding normalizes blood pressure patterns and improves neurovascular control.

The research aims are:

1. To determine the effect of meal timing on blood pressure patterns in middle-aged adults.
2. To determine the effect of meal timing on neurovascular control in middle-aged adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 34 kg/m2
* Non-smoking
* Sedentary or recreationally active
* ≤ 2 Alcoholic drinks per day
* Female subjects: Perimenopausal/Postmenopausal

Exclusion Criteria:

* History or evidence of hepatic, renal, hematological, peripheral vascular disease, or stroke/neurovascular disease, diabetes, uncontrolled hypertension, sleep apnea
* On medications used to treat/manage diseases listed above
* Work overnight shifts
* Clinically diagnosed anxiety or depression
* Pregnant or trying to become pregnant
* Significant surgical history
* Other significant medical conditions at investigator's discretion

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Blood Pressure measured continuously over a period of 24 hour | Continuously over a 24-hour period
  Utilize an ambulatory blood pressure monitor to measure blood pressure values continuously over a 24-hour period.
Neurovascular Control: Change in the brain blood flow | Baseline and 5 weeks
  Change in brain blood flow will be measured using a transcranial Doppler ultrasound in response to a breathing test.
Neurovascular Control: Change in the blood pressure | Baseline and 5 weeks
  Change in blood pressure in response to a breathing test.
Neurovascular Control: change in the sympathetic nerve activity | Baseline and 5 weeks
  Change in sympathetic nerve activity will be measured using microneurography in response to a breathing test.

CONTACTS AND LOCATIONS:
Overall Officials: Jill N Barnes, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ingelsson E, Bjorklund-Bodegard K, Lind L, Arnlov J, Sundstrom J. Diurnal blood pressure pattern and risk of congestive heart failure. JAMA. 2006 Jun 28;295(24):2859-66. doi: 10.1001/jama.295.24.2859. PMID 16804152
- [Background] de la Sierra A, Redon J, Banegas JR, Segura J, Parati G, Gorostidi M, de la Cruz JJ, Sobrino J, Llisterri JL, Alonso J, Vinyoles E, Pallares V, Sarria A, Aranda P, Ruilope LM; Spanish Society of Hypertension Ambulatory Blood Pressure Monitoring Registry Investigators. Prevalence and factors associated with circadian blood pressure patterns in hypertensive patients. Hypertension. 2009 Mar;53(3):466-72. doi: 10.1161/HYPERTENSIONAHA.108.124008. Epub 2009 Jan 26. PMID 19171788
- [Background] Loredo JS, Nelesen R, Ancoli-Israel S, Dimsdale JE. Sleep quality and blood pressure dipping in normal adults. Sleep. 2004 Sep 15;27(6):1097-103. doi: 10.1093/sleep/27.6.1097. PMID 15532203
- [Background] Verdecchia P, Porcellati C, Schillaci G, Borgioni C, Ciucci A, Battistelli M, Guerrieri M, Gatteschi C, Zampi I, Santucci A, Santucci C, Reboldi G, et al. Ambulatory blood pressure. An independent predictor of prognosis in essential hypertension. Hypertension. 1994 Dec;24(6):793-801. doi: 10.1161/01.hyp.24.6.793. PMID 7995639
- [Background] Verdecchia P, Schillaci G, Gatteschi C, Zampi I, Battistelli M, Bartoccini C, Porcellati C. Blunted nocturnal fall in blood pressure in hypertensive women with future cardiovascular morbid events. Circulation. 1993 Sep;88(3):986-92. doi: 10.1161/01.cir.88.3.986. PMID 8353926
- [Background] Hajjar I, Selim M, Novak P, Novak V. The relationship between nighttime dipping in blood pressure and cerebral hemodynamics in nonstroke patients. J Clin Hypertens (Greenwich). 2007 Dec;9(12):929-36. doi: 10.1111/j.1524-6175.2007.07342.x. PMID 18046099
- [Background] Grassi G, Seravalle G, Quarti-Trevano F, Dell'Oro R, Bombelli M, Cuspidi C, Facchetti R, Bolla G, Mancia G. Adrenergic, metabolic, and reflex abnormalities in reverse and extreme dipper hypertensives. Hypertension. 2008 Nov;52(5):925-31. doi: 10.1161/HYPERTENSIONAHA.108.116368. Epub 2008 Sep 8. PMID 18779438
- [Background] Pearson TA, Blair SN, Daniels SR, Eckel RH, Fair JM, Fortmann SP, Franklin BA, Goldstein LB, Greenland P, Grundy SM, Hong Y, Miller NH, Lauer RM, Ockene IS, Sacco RL, Sallis JF Jr, Smith SC Jr, Stone NJ, Taubert KA. AHA Guidelines for Primary Prevention of Cardiovascular Disease and Stroke: 2002 Update: Consensus Panel Guide to Comprehensive Risk Reduction for Adult Patients Without Coronary or Other Atherosclerotic Vascular Diseases. American Heart Association Science Advisory and Coordinating Committee. Circulation. 2002 Jul 16;106(3):388-91. doi: 10.1161/01.cir.0000020190.45892.75. No abstract available. PMID 12119259
- [Background] Douma LG, Gumz ML. Circadian clock-mediated regulation of blood pressure. Free Radic Biol Med. 2018 May 1;119:108-114. doi: 10.1016/j.freeradbiomed.2017.11.024. Epub 2017 Dec 2. PMID 29198725
- [Background] Longo VD, Panda S. Fasting, Circadian Rhythms, and Time-Restricted Feeding in Healthy Lifespan. Cell Metab. 2016 Jun 14;23(6):1048-1059. doi: 10.1016/j.cmet.2016.06.001. PMID 27304506
- [Background] Panda S. Circadian physiology of metabolism. Science. 2016 Nov 25;354(6315):1008-1015. doi: 10.1126/science.aah4967. PMID 27885007
- [Background] Su WL, J. Guo, Z., and Gong, M.C. Time of Food Intake is an Important Determinant of Blood Pressure Circadian Rhythm. Hypertension. 2015;66:AP:225.
- [Background] Nikolaeva S, Pradervand S, Centeno G, Zavadova V, Tokonami N, Maillard M, Bonny O, Firsov D. The circadian clock modulates renal sodium handling. J Am Soc Nephrol. 2012 Jun;23(6):1019-26. doi: 10.1681/ASN.2011080842. Epub 2012 Mar 22. PMID 22440902
- [Background] Grassi G, Bombelli M, Seravalle G, Dell'Oro R, Quarti-Trevano F. Diurnal blood pressure variation and sympathetic activity. Hypertens Res. 2010 May;33(5):381-5. doi: 10.1038/hr.2010.26. Epub 2010 Mar 5. PMID 20203684
- [Background] Fryar CD, Chen TC, Li X. Prevalence of uncontrolled risk factors for cardiovascular disease: United States, 1999-2010. NCHS Data Brief. 2012 Aug;(103):1-8. PMID 23101933
- [Background] Prevention CfDCa. Vital Signs. 2018.
- [Background] Palsson R, Patel UD. Cardiovascular complications of diabetic kidney disease. Adv Chronic Kidney Dis. 2014 May;21(3):273-80. doi: 10.1053/j.ackd.2014.03.003. PMID 24780455
- [Background] Chamberlain JJ, Johnson EL, Leal S, Rhinehart AS, Shubrook JH, Peterson L. Cardiovascular Disease and Risk Management: Review of the American Diabetes Association Standards of Medical Care in Diabetes 2018. Ann Intern Med. 2018 May 1;168(9):640-650. doi: 10.7326/M18-0222. Epub 2018 Apr 3. PMID 29610837
- [Background] Luchsinger JA. Type 2 diabetes, related conditions, in relation and dementia: an opportunity for prevention? J Alzheimers Dis. 2010;20(3):723-36. doi: 10.3233/JAD-2010-091687. PMID 20413862
- [Background] Fagard RH, Celis H, Thijs L, Staessen JA, Clement DL, De Buyzere ML, De Bacquer DA. Daytime and nighttime blood pressure as predictors of death and cause-specific cardiovascular events in hypertension. Hypertension. 2008 Jan;51(1):55-61. doi: 10.1161/HYPERTENSIONAHA.107.100727. Epub 2007 Nov 26. PMID 18039980
- [Background] Boggia J, Li Y, Thijs L, Hansen TW, Kikuya M, Bjorklund-Bodegard K, Richart T, Ohkubo T, Kuznetsova T, Torp-Pedersen C, Lind L, Ibsen H, Imai Y, Wang J, Sandoya E, O'Brien E, Staessen JA; International Database on Ambulatory blood pressure monitoring in relation to Cardiovascular Outcomes (IDACO) investigators. Prognostic accuracy of day versus night ambulatory blood pressure: a cohort study. Lancet. 2007 Oct 6;370(9594):1219-29. doi: 10.1016/S0140-6736(07)61538-4. PMID 17920917
- [Background] Fagard RH, Thijs L, Staessen JA, Clement DL, De Buyzere ML, De Bacquer DA. Night-day blood pressure ratio and dipping pattern as predictors of death and cardiovascular events in hypertension. J Hum Hypertens. 2009 Oct;23(10):645-53. doi: 10.1038/jhh.2009.9. Epub 2009 Feb 19. PMID 19225527
- [Background] Fagard RH, Thijs L, Staessen JA, Clement DL, De Buyzere ML, De Bacquer DA. Prognostic significance of ambulatory blood pressure in hypertensive patients with history of cardiovascular disease. Blood Press Monit. 2008 Dec;13(6):325-32. doi: 10.1097/MBP.0b013e32831054f5. PMID 18756173
- [Background] Mancia G, Bombelli M, Facchetti R, Madotto F, Corrao G, Trevano FQ, Grassi G, Sega R. Long-term prognostic value of blood pressure variability in the general population: results of the Pressioni Arteriose Monitorate e Loro Associazioni Study. Hypertension. 2007 Jun;49(6):1265-70. doi: 10.1161/HYPERTENSIONAHA.107.088708. Epub 2007 Apr 23. PMID 17452502
- [Background] De Nicola L, Conte G, Minutolo R. Prediabetes as a Precursor to Diabetic Kidney Disease. Am J Kidney Dis. 2016 Jun;67(6):817-9. doi: 10.1053/j.ajkd.2016.03.411. No abstract available. PMID 27211364
- [Background] Sorensen BM, Houben AJ, Berendschot TT, Schouten JS, Kroon AA, van der Kallen CJ, Henry RM, Koster A, Sep SJ, Dagnelie PC, Schaper NC, Schram MT, Stehouwer CD. Prediabetes and Type 2 Diabetes Are Associated With Generalized Microvascular Dysfunction: The Maastricht Study. Circulation. 2016 Nov 1;134(18):1339-1352. doi: 10.1161/CIRCULATIONAHA.116.023446. Epub 2016 Sep 27. PMID 27678264
- [Background] Brotman DJ, Davidson MB, Boumitri M, Vidt DG. Impaired diurnal blood pressure variation and all-cause mortality. Am J Hypertens. 2008 Jan;21(1):92-7. doi: 10.1038/ajh.2007.7. PMID 18091750
- [Background] Ohkubo T, Imai Y, Tsuji I, Nagai K, Watanabe N, Minami N, Kato J, Kikuchi N, Nishiyama A, Aihara A, Sekino M, Satoh H, Hisamichi S. Relation between nocturnal decline in blood pressure and mortality. The Ohasama Study. Am J Hypertens. 1997 Nov;10(11):1201-7. doi: 10.1016/s0895-7061(97)00274-4. PMID 9397237
- [Background] Viera AJ, Shimbo D. Ambulatory blood pressure phenotypes and the risk for hypertension. Curr Hypertens Rep. 2014 Oct;16(10):481. doi: 10.1007/s11906-014-0481-5. PMID 25139779
- [Background] Su W, Guo Z, Randall DC, Cassis L, Brown DR, Gong MC. Hypertension and disrupted blood pressure circadian rhythm in type 2 diabetic db/db mice. Am J Physiol Heart Circ Physiol. 2008 Oct;295(4):H1634-41. doi: 10.1152/ajpheart.00257.2008. Epub 2008 Aug 15. PMID 18708447
- [Background] Su W, Xie Z, Guo Z, Duncan MJ, Lutshumba J, Gong MC. Altered clock gene expression and vascular smooth muscle diurnal contractile variations in type 2 diabetic db/db mice. Am J Physiol Heart Circ Physiol. 2012 Feb 1;302(3):H621-33. doi: 10.1152/ajpheart.00825.2011. Epub 2011 Dec 2. PMID 22140039
- [Background] Barr EL, Zimmet PZ, Welborn TA, Jolley D, Magliano DJ, Dunstan DW, Cameron AJ, Dwyer T, Taylor HR, Tonkin AM, Wong TY, McNeil J, Shaw JE. Risk of cardiovascular and all-cause mortality in individuals with diabetes mellitus, impaired fasting glucose, and impaired glucose tolerance: the Australian Diabetes, Obesity, and Lifestyle Study (AusDiab). Circulation. 2007 Jul 10;116(2):151-7. doi: 10.1161/CIRCULATIONAHA.106.685628. Epub 2007 Jun 18. PMID 17576864
- [Background] Gupta AK, Greenway FL, Cornelissen G, Pan W, Halberg F. Prediabetes is associated with abnormal circadian blood pressure variability. J Hum Hypertens. 2008 Sep;22(9):627-33. doi: 10.1038/jhh.2008.32. Epub 2008 May 15. PMID 18480832
- [Background] Oosterman JE, Kalsbeek A, la Fleur SE, Belsham DD. Impact of nutrients on circadian rhythmicity. Am J Physiol Regul Integr Comp Physiol. 2015 Mar 1;308(5):R337-50. doi: 10.1152/ajpregu.00322.2014. Epub 2014 Dec 17. PMID 25519730
- [Background] Chaix A, Zarrinpar A, Miu P, Panda S. Time-restricted feeding is a preventative and therapeutic intervention against diverse nutritional challenges. Cell Metab. 2014 Dec 2;20(6):991-1005. doi: 10.1016/j.cmet.2014.11.001. PMID 25470547
- [Background] Rothschild J, Hoddy KK, Jambazian P, Varady KA. Time-restricted feeding and risk of metabolic disease: a review of human and animal studies. Nutr Rev. 2014 May;72(5):308-18. doi: 10.1111/nure.12104. Epub 2014 Apr 16. PMID 24739093
- [Background] Barnosky AR, Hoddy KK, Unterman TG, Varady KA. Intermittent fasting vs daily calorie restriction for type 2 diabetes prevention: a review of human findings. Transl Res. 2014 Oct;164(4):302-11. doi: 10.1016/j.trsl.2014.05.013. Epub 2014 Jun 12. PMID 24993615
- [Background] Gill S, Le HD, Melkani GC, Panda S. Time-restricted feeding attenuates age-related cardiac decline in Drosophila. Science. 2015 Mar 13;347(6227):1265-9. doi: 10.1126/science.1256682. PMID 25766238
- [Background] Hatori M, Vollmers C, Zarrinpar A, DiTacchio L, Bushong EA, Gill S, Leblanc M, Chaix A, Joens M, Fitzpatrick JA, Ellisman MH, Panda S. Time-restricted feeding without reducing caloric intake prevents metabolic diseases in mice fed a high-fat diet. Cell Metab. 2012 Jun 6;15(6):848-60. doi: 10.1016/j.cmet.2012.04.019. Epub 2012 May 17. PMID 22608008
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Background] Patterson RE, Laughlin GA, LaCroix AZ, Hartman SJ, Natarajan L, Senger CM, Martinez ME, Villasenor A, Sears DD, Marinac CR, Gallo LC. Intermittent Fasting and Human Metabolic Health. J Acad Nutr Diet. 2015 Aug;115(8):1203-12. doi: 10.1016/j.jand.2015.02.018. Epub 2015 Apr 6. No abstract available. PMID 25857868
- [Background] Mager DE, Wan R, Brown M, Cheng A, Wareski P, Abernethy DR, Mattson MP. Caloric restriction and intermittent fasting alter spectral measures of heart rate and blood pressure variability in rats. FASEB J. 2006 Apr;20(6):631-7. doi: 10.1096/fj.05-5263com. PMID 16581971
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2018 May 15;71(19):e127-e248. doi: 10.1016/j.jacc.2017.11.006. Epub 2017 Nov 13. No abstract available. PMID 29146535
- [Background] Rickards CA, Johnson BD, Harvey RE, Convertino VA, Joyner MJ, Barnes JN. Cerebral blood velocity regulation during progressive blood loss compared with lower body negative pressure in humans. J Appl Physiol (1985). 2015 Sep 15;119(6):677-85. doi: 10.1152/japplphysiol.00127.2015. Epub 2015 Jul 2. PMID 26139213
- [Background] Barnes JN. Exercise, cognitive function, and aging. Adv Physiol Educ. 2015 Jun;39(2):55-62. doi: 10.1152/advan.00101.2014. PMID 26031719
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Klempel MC, Kroeger CM, Varady KA. Alternate day fasting (ADF) with a high-fat diet produces similar weight loss and cardio-protection as ADF with a low-fat diet. Metabolism. 2013 Jan;62(1):137-43. doi: 10.1016/j.metabol.2012.07.002. Epub 2012 Aug 11. PMID 22889512
- [Background] Varady KA, Bhutani S, Klempel MC, Kroeger CM, Trepanowski JF, Haus JM, Hoddy KK, Calvo Y. Alternate day fasting for weight loss in normal weight and overweight subjects: a randomized controlled trial. Nutr J. 2013 Nov 12;12(1):146. doi: 10.1186/1475-2891-12-146. PMID 24215592
- [Background] Trepanowski JF, Kroeger CM, Barnosky A, Klempel M, Bhutani S, Hoddy KK, Rood J, Ravussin E, Varady KA. Effects of alternate-day fasting or daily calorie restriction on body composition, fat distribution, and circulating adipokines: Secondary analysis of a randomized controlled trial. Clin Nutr. 2018 Dec;37(6 Pt A):1871-1878. doi: 10.1016/j.clnu.2017.11.018. Epub 2017 Dec 5. PMID 29258678